CLINICAL TRIAL: NCT05181332
Title: Predictive Models of Hepatic Decompensation and Survival Outcomes in Pediatric Patients With Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yuhan Yang, Associate Professor, West China Hospital
Other Study IDs: HX-2021523
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Cirrhosis; Biliary Atresia; Choledochal Cyst; Primary Sclerosing Cholangitis; HBV; HCV; Autoimmune Hepatitis
MeSH Terms: conditions — Fibrosis; Biliary Atresia; Choledochal Cyst; Cholangitis, Sclerosing; Hepatitis, Autoimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: The internal cohort was retrospectively enrolled in West China Hospital, Sichuan University from June 2010 and December 2020. It is a training and internal validation cohort.
  Interventions: Other: Prediction model
- Prospective cohort: The same inclusion/exclusion criteria were applied for the same center prospectively. It is a external validation cohort.
  Interventions: Other: Prediction model

INTERVENTIONS:
Other: Prediction model — Clinical models were developed and validated to predict liver-related complications and survival outcomes in pediatric patients with biopsy-proven with cirrhosis.

SUMMARY:
The aim of this study was to developed and validated models to predict hepatic decompensation and survivals in pediatric patients with cirrhosis and compared these models with currently available models.

DETAILED DESCRIPTION:
Noninvasive liver fibrosis tests such as the NAFLD fibrosis score (NFS), Hepascore, and transient elastography were specifically developed to predict fibrosis and can help predict patients with NAFLD at the highest risk of developing liver-related complications. These tests have been widely applied in adult cirrhosis. The accuracy of these models, however, may be influenced by patient factors including age, body mass index, and diabetes, potentially limiting their prognostic accuracy and clinical practicability in children. Therefore, it is currently unknown how to best predict hepatic decompensation and survival outcomes among pediatric patients with cirrhosis. To fill this knowledge gap, the investigators performed a retrospective-prospective cohort study with the aim of developing and validating a clinical model to predict liver-related complications and survival outcomes in pediatric patients with biopsy-proven with cirrhosis. Secondly, the investigators aimed to compare the predictive accuracy with currently available noninvasive model.

ELIGIBILITY:
Inclusion Criteria:

* Age up to 18 years old
* No previous episodes of clinical decompensation
* With written informed consent

Exclusion Criteria:

* Clinical data missing
* Without written informed consent

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with cirrhosis who were diagnosed histologically with definite pathologic specimens.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Hepatic decompensation | At least 5-year follow up
  The primary outcome was the first event of hepatic decompensation, defined by the occurrence of any of the following: ascites (identified or confirmed by abdominal ultrasound), upper gastrointestinal bleeding secondary to portal hypertension (confirmed by endoscopy in the presence of gastroesophageal varices or portal hypertensive gastropathy), or hepatic encephalopathy (established by clinical parameters, neuropsychological tests, or electroencephalogram)

SECONDARY OUTCOMES:
Overall survival | At least 5-year follow up
  The endpoint was defined as the occurrence of death or the last follow-up. Patients were followed from the day of liver biopsy until the occurrence of death, liver transplant, or last visit. The outcome was evaluated by an experienced hepatologist in each center every 3-6 months. At each visit, a medical history, physical examination, and standard laboratory tests were performed.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No